CLINICAL TRIAL: NCT07071545
Title: Impact of Regular Physical Activity in Normal-Weight Individuals With Type 2 Diabetes and Abdominal Obesity: Nationwide Cohort Study
Brief Title: Effect of Regular Physical Activity in Normal-Weight Individuals With Type 2 Diabetes and Abdominal Obesity
Acronym: PA-NormalWtDM
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ki Hong Choi, Professor, Samsung Medical Center
Other Study IDs: DM_abdominalobesity
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Diabetes (DM); Physical Activity
Keywords: abdominal obesity; physical activity; Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity; Obesity, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Abdominal obesity: Individuals were classified as having abdominal obesity.
  Interventions: Behavioral: Regular physical activity; Behavioral: No regular physical activity
- Without abdominal obesity: Individuals were classified as not having abdominal obesity.

INTERVENTIONS:
Behavioral: Regular physical activity — Moderate-to-vigorous physical activity at least three times per week.
  Groups: Abdominal obesity
Behavioral: No regular physical activity — The group that did not engage in physical activity according to the guidelines
  Groups: Abdominal obesity

SUMMARY:
Individuals with T2DM accompanied by abdominal obesity tend to experience worse clinical outcomes. To identify modifiable factors that may improve these outcomes, the investigators conducted a retrospective cohort study using data from the Korean National Health Insurance Service (K-NHIS) database to evaluate the impact of regular physical activity.

DETAILED DESCRIPTION:
It is well established that patients with T2DM and abdominal obesity have worse clinical outcomes. This holds true even among individuals with a normal body weight but central (abdominal) obesity. In this study, the investigators aimed to determine whether engaging in regular physical activity (defined as vigorous exercise at least three times per week) is associated with improved clinical outcomes in normal-weight individuals with abdominal obesity. Specifically, we compared the incidence of MACCE between normal-weight patients with type 2 diabetes who had abdominal obesity and those who did not.

ELIGIBILITY:
Inclusion Criteria:

- Patients who were newly diagnosed with T2DM and had a normal body weight at the time of diagnosis.

Exclusion Criteria:

* Patients with any pre-existing diabetes-related complications
* Patients who were overweight or obese based on BMI criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were newly diagnosed with T2DM and had a normal body weight at the time of diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 249247 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cerevrovascular events (MACCE) | 10 years after diagnosed T2DM
  Composite of all-cause death, myocardial infarction, ischemic stroke, heart failure

SECONDARY OUTCOMES:
All cause death | 10 years after diagnosed T2DM
  Death from all cause
myocardial infarction | 10 years after diagnosed T2DM
  MI with hospitalization
Ischemic stroke | 10 years after diagnosed T2DM
  Ischemic stroke after diagnosed T2DM
Heart failure | 10 years after diagnosed T2DM
  HF with hospitalization

IPD SHARING:
Plan to Share IPD: Undecided